CLINICAL TRIAL: NCT06427174
Title: Analgesic Efficacy of Us Guided Fascia Iliaca Block Versus Caudal Block in Pediatric Graft Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Atef Ahmed, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FB vs CB
Record Dates: First submitted 2024-05-18; First posted 2024-05-23 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Surgery
Keywords: Fascia iliaca block, analgesia, pediatric surgeries
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patients and anesthesiologist won't know which group is patients will selected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia iliaca group (Active Comparator): For the group who will receive the fascia iliaca block …. After induction of the general anesthesia and before skin incision, fascia iliaca block will be performed in the patient while he is in the supine position after sterilization of skin over the groin area at the side from which split thickness graft will be taken, high frequency ultrasound probe
  Interventions: Drug: Fascia iliaca block
- Caudal block (Active Comparator): And the second group will receive the caudal block, we use bupivacaine 0.5 mg / kg.
  With the patient in the left lateral decubitus position and the hips and knees flexed, the sacral hiatus can be identified .First of all, the posterior superior iliac spines are palpated via anatomical landmarks, the line between both spines (Tuffier's line) representing the base of an equilateral triangle the tip of which indicates the position of the sacral hiatus. The sacrococcygeal ligament can be palpated between the two sacral cornua, which is where the needle should penetrate the skin at an approximate 45° angle. Once the ligament has been passed, a flatter angle is adjusted by descending the needle before it can be advanced to the correct final position.
  Interventions: Drug: Caudal block

INTERVENTIONS:
Drug: Fascia iliaca block — For the group who will receive the fascia iliaca block …. After induction of the general anesthesia and before skin incision, fascia iliaca block will be performed in the patient while he is in the supine position
  Arms: Fascia iliaca group
Drug: Caudal block — second group will receive the caudal block, we use bupivacaine 0.5 mg / kg.
  Arms: Caudal block

SUMMARY:
The study is aimed to determine which of the two methods , either the fascia iliaca block or the caudal block is better in managing the post operative pain and by which decreasing the consumption of analgesic drugs post operatively and making the patient more comfortable.

DETAILED DESCRIPTION:
Split-thickness skin grafting is the current standard of care for the reconstructive procedures in managing burn injuries and traumatic tissue defects. Harvesting split-thickness skin creates a new partial thickness wound that is referred to as the donor site.(1) Donor site pain is one of the most distressing symptoms reported by patients in the early postoperative period.4,5 Larger donor sites stimulate a greater number of pain receptors and consequently pain is proportional to the size of the graft harvested.6 Often, the donor site is reported to be more painful than the recipient site,7 affecting early mobilization, sleep, and need for analgesics postoperatively.(1) Most commonly split thickness auto-grafts are harvested from a convenient and minimally aesthetically intrusive site; often the lateral thigh area, which is innervated by lateral femoral cutaneous nerve (LFCN). However if a larger graft area in needed then it will be obtained from the anterior aspect of the thigh, which is innervated by the femoral nerve.(2) Regional nerve blockade has been proposed for skin graft harvest and proofed to provide better and longer standing analgesia.(2) Application of fascia iliaca compartment block involves the distribution of anesthesia to the territories of the femoral and lateral cutaneous nerves(3) American society of regional anesthesia and pain medicine recommendations on local anesthetics in pediatric regional anesthesia in 2018 stated that the ultrasound guided fascial plane blocks as fascia iliaca block can be successfully and safely performed using a recommended dose of 0.25-0.75 mg/kg of bupivacaine 0.25%.(4) Prolongation of analgesia after any surgery is the goal of any phsyician ,and Fascia Iliaca Block (FIB), which is widely used for postoperative analgesia in many surgeries, is a nerve block technique with proven efficacy. but which has the superior effect of numbing the pain ..Is it the fascia iliaca erve block or the caudal block .

The objective of this study is to compare post operative analgesic effect and safety of fascia iliaca nerve block versus caudal block in pediatric patient undergoing a graft surgery .

ELIGIBILITY:
Inclusion Criteria:

* Age 2- 12 years. ASA I - II Scheduled for split thickness grafting. Availability and suitability of lateral and anterior aspects of the thigh as a donor site.

Exclusion Criteria:

* Patient's gaurdian refusal to participate in the study. Known allergy to local anesthetics Coagulopathy. Patient with motor or sensory deficits in lower extremities. Prior surgery of the inguinal or suprainguinal area . Children who are morbidly obese (BMI≥30) because ultrasound guided regional anesthesia could be too technically difficult.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia using FLACC score | 1-24 hour postiperative
  Postoperative analgesia using FLACC score

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ta Mohamed, Principal Investigator — Lecturer doctor

REFERENCES:
- [Background] Wiegele M, Marhofer P, Lonnqvist PA. Caudal epidural blocks in paediatric patients: a review and practical considerations. Br J Anaesth. 2019 Apr;122(4):509-517. doi: 10.1016/j.bja.2018.11.030. Epub 2019 Feb 1. PMID 30857607
- [Background] Bromage PR. A comparison of the hydrochloride salts of lignocaine and prilocaine for epidural analgesia. Br J Anaesth. 1965 Oct;37(10):753-61. doi: 10.1093/bja/37.10.753. No abstract available. PMID 5847259
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Suresh S, Ecoffey C, Bosenberg A, Lonnqvist PA, de Oliveira GS Jr, de Leon Casasola O, de Andres J, Ivani G. The European Society of Regional Anaesthesia and Pain Therapy/American Society of Regional Anesthesia and Pain Medicine Recommendations on Local Anesthetics and Adjuvants Dosage in Pediatric Regional Anesthesia. Reg Anesth Pain Med. 2018 Feb;43(2):211-216. doi: 10.1097/AAP.0000000000000702. PMID 29319604
- [Background] Shteynberg A, Riina LH, Glickman LT, Meringolo JN, Simpson RL. Ultrasound guided lateral femoral cutaneous nerve (LFCN) block: safe and simple anesthesia for harvesting skin grafts. Burns. 2013 Feb;39(1):146-9. doi: 10.1016/j.burns.2012.02.015. Epub 2012 May 30. PMID 22657583
- [Background] Shank ES, Martyn JA, Donelan MB, Perrone A, Firth PG, Driscoll DN. Ultrasound-Guided Regional Anesthesia for Pediatric Burn Reconstructive Surgery: A Prospective Study. J Burn Care Res. 2016 May-Jun;37(3):e213-7. doi: 10.1097/BCR.0000000000000174. PMID 25412051
- [Background] Sinha S, Schreiner AJ, Biernaskie J, Nickerson D, Gabriel VA. Treating pain on skin graft donor sites: Review and clinical recommendations. J Trauma Acute Care Surg. 2017 Nov;83(5):954-964. doi: 10.1097/TA.0000000000001615. PMID 28598907